CLINICAL TRIAL: NCT03607994
Title: Randomized Controlled Pilot Trial of HIRREM-SOP for Insomnia
Brief Title: Study of the Effects of HIRREM-SOP for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00051980
Record Dates: First submitted 2018-07-13; First posted 2018-07-31 (Actual); Results first posted 2021-06-22 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-05

CONDITIONS: Insomnia; Sleep Deprivation
Keywords: Neurotechnology; Autonomic Dysregulation; Hyperarousal; Brain Electrical Activity; Closed-loop; Acoustic Stimulation; Allostasis; Insomnia; HIRREM-SOP; Sleep Deprivation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Deprivation; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: This study will compare acoustic stimulation linked to brainwave activity (HIRREM-SOP, along with continued current care, BCC) with acoustic stimulation not linked to brainwave activity (NCC, along with continued current care). The participants in the NCC group with will offered the opportunity to crossover and receive a course of BCC at the end of their original participation.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- HIRREM-SOP (BCC (Active Comparator): Acoustic stimulation linked to brainwave activity and continued current care.
  Interventions: Device: HIRREM-SOP
- nonspecific acoustic stimulation (NCC) (Other): Continued current care and acoustic stimulation that is not linked to brainwave activity.
  Interventions: Device: HIRREM-SOP; Device: NCC

INTERVENTIONS:
Device: HIRREM-SOP — HIRREM-SOP is an updated version of HIRREM. It is a novel, noninvasive, closed-loop, brainwave mirroring, acoustic stimulation neurotechnology to support relaxation and auto-calibration of neural oscillations, using auditory tones to reflect brain frequencies in near real time.
Device: NCC — Nonspecific acoustic stimulation with randomly generated tones not linked to brain activity.
  Arms: nonspecific acoustic stimulation (NCC)

SUMMARY:
Prior research studies have shown benefit for use of a technique called High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM®), to reduce symptoms of moderate to severe insomnia. HIRREM uses scalp sensors to monitor brain electrical activity, and software algorithms translate selected brain frequencies into audible tones in real time. Those tones (acoustic stimulation) are reflected back to participants via ear buds in as little as four milliseconds, providing the brain an opportunity to self-adjust and balance its electrical pattern.

The purpose of this research study is to determine the effects of HIRREM-SOP, an updated version of this technology that is based on the HIRREM approach, but now includes new hardware and software, a standardized series of HIRREM protocols, and a fixed number of sessions. Adults over the age of 18 who have documented sleep trouble that place them in the category of subthreshold (mild), moderate, or severe clinical insomnia as defined by the Insomnia Severity Index, are eligible to participate in the study.

DETAILED DESCRIPTION:
High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM®) is a closed-loop, allostatic, acoustic stimulation neurotechnology that uses software-guided algorithmic analysis to identify and translate selected brain frequencies into audible tones to support real-time self-optimization of brain activity. Prior research demonstrates that the use of HIRREM is associated with reduced symptoms of insomnia, and traumatic stress and anxiety, and improved autonomic cardiovascular regulation across heterogeneous cohorts. HIRREM has been safe and well tolerated in about 500 people across six IRB-approved studies. However, the current in-office HIRREM approach remains very operator dependent (extensive Technologist education and experience) and takes a sizeable time commitment from the participant (typically ten or more sessions of 90-120 minutes each). To reduce participant time required, and operator dependence, while increasing scalability, a new generation of hardware and software has been developed. While based on the same core technology and algorithms to mirror brainwaves with audible tones, this includes the use of faster, 64-bit processing architecture for faster feedback, the use of 4 sensors, and the use of standard protocols, all done with eyes closed (HIRREM-SOP). Although only 2 sensors are active at a time, applying 4 sensors, for which the software can switch from one pair to the other automatically, cuts in half the number of sensor placement changes needed, with reduced session time and interruptions. A modified placebo condition now includes random timing and pitch of the tones, which have not been acoustically engineered. This pilot study will evaluate feasibility of this standardized, enhanced approach, and the effectiveness of blinding for the placebo condition in participants with symptoms of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Insomnia (Insomnia Severity Index ≥ 8) persisting by self-report for at least a month
* Subjects must have the ability to comply with basic instructions and be able to comfortably sit still with the sensor leads attached

Exclusion Criteria:

* Unable, unwilling, or incompetent to provide informed consent
* Physically unable to come to the study visits, or to sit in a chair for several hours
* Known seizure disorder
* Known obstructive sleep apnea
* Diagnosed periodic limb movement disorder or known restless legs syndrome
* Known urinary problem (i.e. benign prostatic hypertrophy) which is the likely cause of the sleep disturbance
* Severe hearing impairment (because the subject will be using ear buds during HIRREM-SOP)
* Ongoing need for treatment with opiate, benzodiazepine, or anti-psychotic medications, anti-depressant medications (SSRI, or SNRI's), sleep medications such as zolpidem or eszopiclone, stimulants such as Adderall, Provigil, or Ritalin, or thyroid hormone
* Anticipated and ongoing use of recreational drugs, alcohol, or energy drinks
* Weight is over the chair limit (285 pounds)
* Currently in another active intervention research study
* Previous history of receiving or using HIRREM, BWO, HIRREM-SOP, or the wearable B2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Tegeler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Department of Neurology, Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HIRREM-SOP (BCC): Acoustic stimulation linked to brainwave activity and continued current care.
  HIRREM-SOP: HIRREM-SOP is an updated version of HIRREM. It is a novel, noninvasive, closed-loop, brainwave mirroring, acoustic stimulation neurotechnology to support relaxation and auto-calibration of neural oscillations, using auditory tones to reflect brain frequencies in near real time.
Period: Overall Study
Arm/Group | HIRREM-SOP (BCC) | Nonspecific Acoustic Stimulation (NCC)
Started | 10 | 12
Completed | 9 | 11
Not Completed | 1 | 1
Not completed — Discontinued intervention (started sessions and dropped out due to time commitment and schedule) | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIRREM-SOP (BCC) | Nonspecific Acoustic Stimulation (NCC) | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (7.96) | 54.67 (19.19) | 56.45 (14.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — The ISI is a 7 question, self-reported measure to evaluate symptoms of insomnia, with responses from 0-4 for each question, yielding scores ranging from 0-28. Lower scores represent better outcomes. The primary outcome will be change from enrollment to 4-6 weeks after completion of the intervention.
  units on a scale | 14.90 (4.65) | 18.00 (3.07) | 16.59 (4.09)
Duration with Sleep Trouble [Mean (Standard Deviation); unit: years] | 8.98 (11.43) | 5.28 (3.89) | 6.96 (8.22)

OUTCOME MEASURES:

1. Primary Outcome: Change in ISI Score From V1 to V3
Description: The severity of insomnia symptoms is measured using the ISI with each data collection visit. The ISI is a 7 question measure, with responses from 0-4 for each question, yielding scores ranging from 0-28. Higher scores indicate the strength of the insomnia severity.
Time Frame: Baseline, V2 (0-14 days after intervention completion), V3 (4-6 weeks following V2)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HIRREM-SOP (BCC) | Nonspecific Acoustic Stimulation (NCC)
Number analyzed (Participants) | 10 | 12
score on a scale | -7.27 (1.55) | -4.69 (1.40)

2. Secondary Outcome: Number of Participants That Believe They Are Receiving HIRREM-SOP
Description: The participant will indicate which arm of the intervention they believe they are receiving. The effectiveness will be evaluated based on the expectation measure regarding group assignment prior to the 5th session.
Time Frame: Baseline, before Session 5, V2 (0-14 days after intervention completion), V3 (4-6 weeks following V2)
Measure: Count of Participants; unit: Participants
Arm/Group | HIRREM-SOP (BCC) | Nonspecific Acoustic Stimulation (NCC)
Number analyzed (Participants) | 10 | 11
Participants
  Guessed BCC Group (Before Session 5) | 7 | 5
  Guessed NCC Group (Before Session 5) | 3 | 6

ADVERSE EVENTS:
Time Frame: 16-18 weeks after completion of the intervention.
Description: No adverse events or serious adverse events documented during study. Participant ST06 did mention unusual symptoms that was documented, but unsure if study related due to stopping meditation and marijuana use, which were both daily occurrences, as well as a diet change. ST06 reported that she does not feel that the sessions caused her issues.
Arm/Group | HIRREM-SOP (BCC) | Nonspecific Acoustic Stimulation (NCC)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 1/10 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIRREM-SOP (BCC) (N=10) | Nonspecific Acoustic Stimulation (NCC) (N=12)
Other (Nervous system disorders) | 1 (1) | 0 (0) — Reported "constant whooshing in ears, pulse in the 80's, and increased hot flashes." ST06 stopping meditation and marijuana use, both daily occurrences, as well as diet change. ST06 stated she did not feel that the sessions caused her issues.

LIMITATIONS AND CAVEATS:
As a pilot study, small sample size was the key limiting factor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT03607994/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT03607994/ICF_001.pdf